CLINICAL TRIAL: NCT04369547
Title: A Double-blind Placebo-controlled Crossover Study of Roflumilast Synaptic Plasticity Enhancement: a TMS-EEG Study
Brief Title: Roflumilast TMS-EEG Plasticity
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Resource limitations
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Alexander McGirr, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REB20-0196
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Synaptic Plasticity
Keywords: rTMS; EEG; Augmented Plasticity
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast (Experimental): Participants will ingest a capsule containing 250mcg of the phosphodiesterase-4 inhibitor roflumilast. Their baseline TMS evoked potentials (TEP) will be recorded over 100 single TMS pulses prior to receiving theta-burst stimulation (TBS; a patterned stimulation) to the left dorsolateral prefrontal cortex (DLPFC). TEP will then be re-recorded at 10, 20, and 30 minutes post-stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation; Drug: Roflumilast
- Placebo (Placebo Comparator): Participants will ingest a capsule identical to that containing the study medication, however, this capsule will be contain a placebo. Their baseline TEP will be recorded over 100 single TMS pulses prior to receiving TBS to the left DLPFC. TEP will then be re-recorded at 10, 20, and 30 minutes post-stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation; Drug: Placebo oral tablet

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Single-pulse transcranial magnetic stimulation and theta-burst stimulation.
Drug: Roflumilast — Roflumilast 250mcg
  Arms: Roflumilast
Drug: Placebo oral tablet — Placebo capsule matched to roflumilast capsule
  Arms: Placebo

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) uses a magnetic field to non-invasively induce electrical function within the brain. Stimulation allows brain cells to change the way that they adapt and communicate with each other, known as 'synaptic plasticity'. It is thought that alterations in these adaptive brain changes underlie the ability of rTMS to treat mental illnesses like depression. rTMS is a Health Canada approved treatment for depression, however, 2/3rds of people fail to show meaningful improvement. This highlights the need for more effective therapeutic means. The purpose of the present study is to augment the therapeutic abilities of rTMS through the conjunctive use of a medication that also increases synaptic plasticity. We will pair TMS with an electroencephalograph (EEG) to measure activity dependent changes in the frontal cortex following rTMS.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, crossover trial will enroll 20 healthy participants. In one arm of the study, participants will randomly receive either 250mcg of roflumilast (a phosphodiesterase-4 inhibitor), or a placebo capsule, and participants will receive the other intervention one week later.

1. The investigators will recruit 20 healthy participants through community advertisement, carefully screened for exclusion factors related to rTMS and roflumilast.
2. Participants will be randomly assigned by random number sequence with allocation concealment to one of two first arms of the crossover study: a) placebo-roflumilast 250mcg and b) roflumilast 250mcg-placebo.
3. Participants will complete the QIDS-SR (Quick Inventory of Depressive Symptoms-Self Report), the BAI (Beck Anxiety Inventory), and the STAI (State Trait Anxiety Inventory).

   Participants will report their perception of physical symptoms (potential side effects) in the 7 days before participating in the study taking the randomized capsule (Toronto Side Effects Scale - 1 Week).
4. Participants will take their blinded capsule at least 30 minutes prior to TBS (theta-burst stimulation).
5. The resting motor threshold of participants will be determined using electromyographic electrodes (EMG). EMG electrodes will be positioned over the first dorsal interosseous (FDI) muscle on the right hand. These electrodes are non-invasive and use an adhesive to stick to the skin.
6. The M1 hand strip will be localized using single pulse TMS (MagPro X100) in conjunction with neuronavigation and an atlas brain.
7. Muscle activation in response to TMS will be measured through motor evoked potentials (MEP). The strength of MEPs in response to differing strengths of single pulse TMS will be used to determine a participants resting motor threshold (RMT). The RMT is the lowest TMS setting at which the FDI muscle responds to TMS stimulus. 80% of the RMT will then be the strength at which TBS protocol will be applied to the DLPFC.
8. Two baselines of TMS Evoked Potentials (TEPs) will be collected via one hundred single-pulse (120% RMT), 0.25Hz) over the F3 site. Each baseline will occur 10 minutes apart.
9. TBS-rTMS will be applied to the DLPFC site. TBS consists of 2s trains every 10s. Each train is composed of 3 pulses at 50Hz, 200ms intervals given at 80% RMT. The total time for this treatment stimulus is 600 pulses over 190s.
10. Following TBS, one hundred TEPs over the F3 site will again be acquired at 10, 20, and 30 minutes after treatment (single pulse, 120%RMT, 0.25Hz).

As this is a cross-over study, participants will return 1 week later to repeat the second arm of the protocol (steps 3-10).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals (no chronic medical conditions).
2. Aged 18-60 years.

Exclusion Criteria:

1. Pregnancy
2. Lactation
3. Epilepsy
4. Previous stroke
5. Current Renal Disease
6. Current Liver Disease
7. Allergy to roflumilast or any of its non-medicinal ingredients
8. Current psychiatric concerns
9. Currently taking any medications that interact with roflumilast
10. Intracranial metallic objects (dental hardware is not an exclusionary criterion)
11. Substance use disorder
12. The inability to refrain from alcohol use for 24 hours prior to stimulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
TMS Evoked Potential amplitude | Baseline versus 10, 20, and 30 minutes following theta-burst stimulation.
  Change in the electrical response of neurons in the dorsolateral prefrontal cortex will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of individual participant data.